CLINICAL TRIAL: NCT06126913
Title: Achieving HIV Viral Suppression in Refugee Settlements in Uganda With Head StART: A Cluster Randomized Trial Evaluating the Effectiveness of Community ART Delivery for People Newly Diagnosed With HIV
Brief Title: HeadStART: Evaluating the Effectiveness of Community ART Delivery for People Newly Diagnosed With HIV
Acronym: HeadStART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelli O'Laughlin, Associate Professor, Departments of Emergency Medicine and Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00016473; R01MH130216 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-11-13 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections; Hiv
Keywords: community ART delivery; HIV; Antiretroviral therapy; Uganda; refugee; humanitarian
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): At sites randomized to standard care, participants newly diagnosed will receive facility-based care per Uganda Ministry of Health (MoH) protocols
- Community Antiretroviral Therapy (Experimental): Newly diagnosed individuals (diagnosed in the prior 6 months) at intervention sites will be offered community ART delivery on a rolling basis during the enrollment window, initiating individuals into groups as close to their date of diagnosis as possible. Newly enrolled individuals will join existing community ART delivery groups, or when a new group is needed based on group size or geographic location, a new group will be formed.
  Interventions: Other: Community Antiretroviral Therapy

INTERVENTIONS:
Other: Community Antiretroviral Therapy — Newly diagnosed individuals (diagnosed in the prior 6 months) at intervention sites will be offered community ART delivery on a rolling basis during the enrollment window, initiating individuals into groups as close to their date of diagnosis as possible. Newly enrolled individuals will join existing community ART delivery groups, or when a new group is needed based on group size or geographic location, a new group will be formed.
  Arms: Community Antiretroviral Therapy

SUMMARY:
This is a cluster randomized controlled trial at 12 health centers in refugee settlements in Uganda aiming to evaluate effectiveness of expansion of community antiretroviral therapy (ART) delivery to people newly diagnosed with HIV in achieving HIV viral suppression.

DETAILED DESCRIPTION:
Community antiretroviral therapy (ART) delivery is a differentiated care model that fosters social support and reduces time and transportation barriers yielding improved engagement in HIV care. In Uganda, to participate in community ART delivery, clients must be "stable" in care (> 1 year on ART and viral load < 1,000 copies/mL). Therefore, persons newly diagnosed with HIV are not eligible for community ART delivery. Community ART delivery may benefit persons newly diagnosed with HIV in refugee settlements by bolstering social support and by bringing ART closer to individuals living in these expansive rural settlements. The primary objective of this research is to evaluate the effectiveness of expanding community ART delivery to clients newly diagnosed with HIV.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Adult ≥18 years of age or mature minors or emancipated minor. Mature minors are defined as individuals 14-17 years of age who have drug or alcohol dependency or a sexually transmitted infection. Emancipated minors are defined as individuals below the age of majority (18 years) who are pregnant, married, have a child, or are self-sufficient.
4. Tested HIV positive in the past 6 months and not already known to be HIV positive.
5. Able to communicate in one of the following 5 study languages: Kiswahili, Runyankore, Kinyarwanda, Somali, or English.

Inclusion criteria for data abstraction only:

1. Adult ≥18 years of age or mature minors or emancipated minor.
2. Tested HIV positive in the past 6 months and not already known to be HIV positive.

Exclusion Criteria:

1. Pregnant and breastfeeding women.
2. Clients deemed by the clinician(s) unfit for community-based care secondary to medical need.
3. Concurrently enrolled in another biomedical clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2720 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
HIV viral suppression at 12 months | 12 months (+/- 2 months)
  HIV viral suppression is defined as <1,000 copies/mL

SECONDARY OUTCOMES:
HIV viral suppression at 6 months | 6 months (+/- 2 months)
  HIV viral suppression is defined as <1,000 copies/mL
Antiretroviral therapy adherence among those virally unsuppressed at 12 months | 12 months (+/- 2 months)
  assessed by determining tenofovir diphosphate blood concentrations among those virally unsuppressed

CONTACTS AND LOCATIONS:
Overall Officials: Kelli N. O'Laughlin, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Diseases Institute, Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT06126913/Prot_SAP_000.pdf